CLINICAL TRIAL: NCT03311737
Title: Compare the Analgesic Effect of Different Anesthesia and Postoperative Analgesic Methods in Uniportal VATS Lung Surgery
Acronym: CDAAMIUVLS
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shanghai Zhongshan Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: zs20170511
Record Dates: First submitted 2017-09-23; First posted 2017-10-17 (Actual); Last update posted 2017-10-17 (Actual); Status verified 2017-09

CONDITIONS: Postoperative Pain; Single-incision Thoracoscopic Surgery
MeSH Terms: conditions — Pain, Postoperative | interventions — Anesthesia, General; Anesthesia, Epidural

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- general anesthesia group (Experimental): The patients in this group receive general anesthesia preoperatively, and use patient controlled intravenous analgesia postoperatively.
  Interventions: Combination Product: general anesthesia
- epidural group (Active Comparator): The patients in this group receive general anesthesia combined with epidural anesthesia, and use patient controlled epidural analgesia postoperatively.
  Interventions: Combination Product: epidural anesthesia

INTERVENTIONS:
Combination Product: general anesthesia — The investigators used general anesthesia preoperatively in uniportal VATS lung surgery
  Arms: general anesthesia group
Combination Product: epidural anesthesia — The investigators used general anesthesia combined with epidural anesthesia preoperatively in uniportal VATS lung surgery
  Arms: epidural group

SUMMARY:
This is a single center, randomized, single blind study to compare the analgesic effect of different anesthesia and postoperative analgesic methods in uniportal VATS lung surgery.

DETAILED DESCRIPTION:
Combining epidural with general anesthesia is regarded as the gold standard of general thoracic surgery. The uniportal VATS lung surgery have advantages of minimal invasive surgical incision, less postoperative pain, and so on. Whether general anesthesia can become an alternative method of combining epidural with general anesthesia in uniportal VATS lung surgery, investigators thus plan to make a comparison on intraoperative stress response, postoperative pain, immune function of patients，and hospital expenses.

ELIGIBILITY:
Inclusion Criteria:

* Patients elective uniportal VATS lung surgery;
* BMI 18-30 kg/m2.

Exclusion Criteria:

* Patient refuse;
* ASA≥3;
* Patients allergic to use anesthetics (propofol,rocuronium), patients with liver and/or kidney and/or mental dysfunction.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2017-09-19 (Actual); Primary Completion 2018-03-31 (Estimated); Study Completion 2018-03-31 (Estimated)

PRIMARY OUTCOMES:
visual analogue scale（VAS） | 1 year
  This scale mainly reflects the patient's pain

CONTACTS AND LOCATIONS:
Locations (1):
- Zhongshan Hospital, Shanghai, Shanghai Municipality, China